CLINICAL TRIAL: NCT04042623
Title: An Open-Label Phase 2a Study to Evaluate the Safety and Efficacy of AVB-S6-500 in Patients With IgA Nephropathy
Brief Title: Study of Safety and Efficacy of AVB-S6-500 in Patients With IgA Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVB500-IGA-001
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: IgA Nephropathy
Keywords: IgAN; AXL inhibitor; Berger's Disease; Proteinuria; Kidney Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with AVB-S6-500 (Experimental): Patients will receive AVB-S6-500 by intravenous infusion every 2 weeks for total of 6 doses.
  Interventions: Drug: AVB-S6-500

INTERVENTIONS:
Drug: AVB-S6-500 — AVB-S6-500 is experimental drug

SUMMARY:
This is an open-label Phase 2a clinical study designed to evaluate the safety and efficacy of AVB-S6-500 in patients with IgA Nephropathy (IgAN). Approximately 24 patients will be enrolled. Several dose levels of AVB-S6-500 may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biopsy-proven IgAN
* Proteinuria ≥ 1g to 3g/24hr
* Stable estimated glomerular filtration rate (eGFR) for at least 3 months prior to screening and ≥ 45 mL/min per 1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration formula
* Systolic BP lesser than or equal to 150 mmHg and diastolic BP lesser than or equal to 100 mmHg
* Patients who have been on a steady dose of ACE or ARB inhibitors for at least 3 months and throughout screening and who are not expected to have their dose adjusted during the study are allowed on study (patients who are not on ACEi/ARB due to inability to tolerate these therapies are also allowed)
* If a sexually-active patient, must agree to use a reliable method of birth control from at least 4 weeks prior to first dose of study drug, during the study and for 1 month following completion of therapy.

Exclusion Criteria:

* Patients with chronic urinary tract infections (UTIs) or taking prophylactic antibiotics to prevent recurrent UTIs
* Treatment with systemic immunosuppressants, including corticosteroids, within 8 weeks of the first dose of study drug
* Rapidly progressing nephropathy defined as falling GFR (≥ 15%) over past 3 mos
* Clinical or biological evidence of diabetes mellitus, systemic lupus erythematosus, IgA vasculitis (Henoch-Schonlein purpura), secondary IgAN, or other renal disease
* Hemoglobin < 9.0 g/dL
* History or clinical evidence of cirrhosis, or liver disease with serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3x upper limit of normal
* Organ transplant recipient (including bone marrow) or a planned transplant during the study
* Have a diagnosis of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection, or positive serology at screening
* Recent active infection requiring hospitalization or i.v. treatment within 30 days prior to the first dose of study drug
* Received transfusion, plasmapheresis or plasma exchange, IV immunoglobulin (IVIg) within 90 days prior to screening
* Malignancy within the past 5 years. Exceptions are squamous cell carcinoma of skin, basal cell carcinoma of skin, and cervical carcinoma in situ which have been excised and are considered cured
* Females who are nursing, pregnant, or intending to become pregnant during the time of the study, or who have a positive pregnancy test at baseline
* Exposure to an investigational drug or device within 90 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
* Known sensitivity to any of the products to be administered during dosing
* Subject will not be available for follow-up assessment
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Prior exposure to AVB-S6-500

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Desir, Study Director — Aravive, Inc.
Locations (2):
- Moonshine Clinical Research, Doral, Florida, United States
- Institute of Nephrology National Academy of Medical Science Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With AVB-S6-500: The subject received a single dose of AVB-S6-500 at 10 mg/kg (total dose 670 mg)
Period: Overall Study
Arm/Group | Treatment With AVB-S6-500
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ukraine | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: Measured by the number of patients with AEs
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: The Effect of AVB-S6-500 on Change From Baseline to End of Treatment in 24-hour Urine Protein Excretion (UPE) in g/Day.
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

3. Primary Outcome: The Effect of AVB-S6-500 on Change From Baseline to End of Treatment in 24-hour Urine Protein Excretion (UPE) in g/Day in the Subset of Patients With Baseline High Proteinuria.
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

4. Primary Outcome: The Effect of AVB-S6-500 on Proportion of Patients With Urinary Protein Equivalent of < 1 g/24 Hours at End of Treatment
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

5. Primary Outcome: The Effect of AVB-S6-500 on Proportion of Patients Who Had at Least a Decrease of 0.5 g/Day Proteinuria From Baseline to End of Treatment.
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

6. Primary Outcome: The Effect of AVB-S6-500 on Change From Baseline to End of Treatment in Urine Albumin/Creatinine Ratios (uACRs).
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

7. Primary Outcome: The Effect of AVB-S6-500 on Change From Baseline to End of Treatment in Estimated Glomerular Filtration Rate (eGFR).
Time Frame: 12 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of Anti-drug Antibody (ADA)
Description: The number of participants with anti-AVB-S6-500 antibodies
Time Frame: 14 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

9. Secondary Outcome: Titers of Anti-AVB-S6-500 Antibodies
Time Frame: 14 weeks
Population: The subject discontinued the study before data were collected, hence the outcome measure was not analyzed.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

10. Secondary Outcome: Apparent Terminal Half-life (t1/2) of AVB-S6-500
Time Frame: 12 weeks
Population: Samples were not analyzed because the study was terminated by the Sponsor.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration of AVB-S6-500 (Cmax)
Time Frame: 12 weeks
Population: Samples were not analyzed because the study was terminated by the Sponsor.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

12. Secondary Outcome: Area Under Time-concentration Curve (AUC)
Time Frame: 12 weeks
Population: Samples were not analyzed because the study was terminated by the Sponsor.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

13. Secondary Outcome: Time of Maximum Observed AVB-S6-500 Concentration (Tmax)
Time Frame: 12 weeks
Population: Samples were not analyzed because the study was terminated by the Sponsor.
Arm/Group | Treatment With AVB-S6-500
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The adverse events data were collected over 1 month period: the subject consented to participate in this study on 11-Feb-2020. On 12-Mar-2020, AVB-S6-500 10 mg/kg (total dose 670 mg) was administered intravenously . The subject did not receive any subsequent doses of AVB-S6-500, nor did she complete the study. The subject underwent post-treatment assessments through telephone contact, as in-person visits were limited due to COVID. The date of early study discontinuation is noted as 06-Apr-2020.
Arm/Group | Treatment With AVB-S6-500
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With AVB-S6-500 (N=1)
Decreased blood pressure (Vascular disorders) | 1 (1)
Rigor (General disorders) | 1 (1)
Feeling heavy (heaviness) in the back (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
After enrollment of one subject, the study was paused due to the COVID-19 pandemic. Subsequently, the sponsor terminated the study due to a change in sponsor priorities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld. However, since the study was terminated, there are no results to be published.

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04042623/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04042623/SAP_001.pdf